CLINICAL TRIAL: NCT04757506
Title: An Investigation of the Effects of Opioid Receptor Blockade on Changes in Self-esteem and Attentional Bias Toward Social Cues
Brief Title: An Investigation of the Effects of Opioid Receptor Blockade on Changes in Self-esteem and Social Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Jennifer Bartz, Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A02-B12-11B
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Self Esteem
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): cellulose-filled capsule
  Interventions: Drug: Placebo
- Naltrexone (Experimental): single 50 mg oral dose naltrexone (capsule)
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — opioid receptor antagonist
  Arms: Naltrexone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the effects of endogenous opioids on self-esteem and attentional bias toward social cues. This is achieved by administering the drug naltrexone, which temporarily decreases endogenous opioid activity.

ELIGIBILITY:
Inclusion Criteria:

* good physical health,
* normal kidney and liver function results from within previous year

Exclusion Criteria:

* allergy to naltrexone
* kidney or liver injury or disorder
* bipolar, panic, or psychotic disorders
* epilepsy
* smoking more than 15 cigarettes per day
* pregnancy
* substance abuse
* use of opioid analgesics, cocaine, recreational drugs (e.g., marijuana, LSD, ecstasy, etc.), or prescription medication (except oral contraceptives) within the past 10 days
* use of over-the-counter drugs (e.g., analgesics, anti-inflammatories, sleeping aids, etc.) or alcohol within the past 24 hours
* current experience of pain (e.g., headache)
* use of anti-diarrheal medications in the 7 days prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-07-09 (Actual); Primary Completion 2013-03-15 (Actual); Study Completion 2013-03-15 (Actual)

PRIMARY OUTCOMES:
Self-esteem | Approximately 2 hours post placebo/drug administration
  Self-reported levels of self-esteem assessed using the Rosenberg Self-Esteem Scale (Rosenberg, 1965). Possible scores range from 1 to 4. Higher scores indicate higher levels of self-esteem.
Attentional bias scores for positive social cues on visual probe task | Approximately 2 hours post placebo/drug administration
  Attentional bias was assessed using a Visual Probe Task. The investigators used a version of the VPT (DeWall, Maner, & Rouby, 2009) designed to assess attentional bias to cues of social acceptance (i.e., smiles). The outcome measure was attentional bias scores, calculated by subtracting mean reaction time scores on "valid" trials from mean reaction time on "invalid" trials. Higher positive scores indicate greater attentional bias to accepting faces.

SECONDARY OUTCOMES:
Attentional bias scores for negative social cues on visual probe task | Approximately 2 hours post placebo/drug administration
  Attentional bias was assessed using a Visual Probe Task. The investigators used a version of the VPT (DeWall, Maner, & Rouby, 2009) designed to assess attentional bias to cues of social rejection (i.e., disapproving faces). The outcome measure was attentional bias scores, calculated by subtracting mean reaction time scores on "valid" trials from mean reaction time on "invalid" trials. Higher positive scores indicate greater attentional bias to disapproving faces.
Reaction times on neutral-neutral trials on visual probe task | Approximately 2 hours post placebo/drug administration
  Reaction times on neutral-neutral trials on the visual probe task were used to assess potential psychomotor side-effects of naltrexone
Self-liking | Approximately 2 hours post placebo/drug administration
  For exploratory purposes, the self-esteem measure (Rosenberg, 1965) was split into two separate subscales examining feelings of self-liking and self-competence as in Tafarodi & Milne, 2002. Self-liking is thought to be more relationally derived and based on internalized perceptions of social approval. Scores range from 1 to 4, with higher scores indicating higher levels of self-liking.
Self-competence | Approximately 2 hours post placebo/drug administration
  For exploratory purposes, the self-esteem measure (Rosenberg, 1965) was split into two separate subscales examining feelings of self-liking and self-competence as in Tafarodi & Milne, 2002. Self-competence is thought to be more autonomously derived and based on past goal pursuit. Scores range from 1 to 4, with higher scores indicating higher levels of self-competence.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bartz, PhD, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available via OSF upon publication of the paper.
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT04757506/Prot_SAP_000.pdf